CLINICAL TRIAL: NCT02593812
Title: The Impact of Standard Medical Care (Dopamine) and Practice on Postural Motor Learning in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: American Parkinson's Disease Association, Inc (Other)
Responsible Party: Principal Investigator, Serene Paul, Postdoctoral Research Associate, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB_00085073
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Parkinson Disease
Keywords: Learning; Practice
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Training "off" medication (Experimental): Participants will train on the postural stepping task before taking their first daily dose of standard Parkinson's medication (dopamine), i.e. while "off" dopamine replacement medication
  Interventions: Behavioral: Stepping training
- Training "on" medication (Other): Participants will train on the postural stepping task after taking their first daily dose of standard Parkinson's medication (dopamine), i.e. while "on" dopamine replacement medication
  Interventions: Behavioral: Stepping training

INTERVENTIONS:
Behavioral: Stepping training — Participants will step rapidly to one of four cued targets. Each trial will consist of 24 steps. Participants will perform 6 blocks of 6 trials per day for 3 consecutive days.

SUMMARY:
The study determines whether standard medical care (dopamine) affects learning and retention of a postural stepping task in people with Parkinson's disease (PD) and whether training on a postural stepping task generalises to performance on an untrained postural task. Half the participants will train on the stepping task after they have taken their first dose of dopamine for the day (i.e. "on" medication state) while the other half will train on the same stepping task before taking their first daily dose of dopamine (i.e. "off" medication state).

DETAILED DESCRIPTION:
Motor learning is critical for acquiring new skills and adapting behaviour, therefore the success of rehabilitation depends on successful motor learning through practice. Motor learning involves the basal ganglia, including both the associative and sensorimotor striatum. Although people with PD are capable of motor learning, they are less efficient and do not achieve the same extent of skill acquisition and retention as people without neurological deficit.

Reductions in endogenous dopamine and reduced dopamine binding associated with loss of dopaminergic receptors due to disease progression may impair motor learning in people with PD. Conflicting evidence suggests that impaired motor learning in PD is due on the one hand to the absence of dopamine but on the other hand to "overdosing" of the basal ganglia with dopamine replacement therapy which suppresses activation of the associative striatum during the early acquisition stages of motor learning.

Understanding which factors improve or degrade motor learning of tasks will allow rehabilitation parameters to be adjusted around standard medical care in order to optimize learning and improve the efficacy of exercise interventions for people with PD. In particular, successful learning of postural tasks that challenge stability may in turn reduce falls.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease confirmed by neurologist
* Hoehn and Yahr stages 1 to 3
* On a stable dose of antiparkinsonian medication for the past month and will continue on this regime for at least another subsequent month
* Walks unaided

Exclusion Criteria:

* Not taking dopamine replacement therapy
* With prior surgical management for PD (e.g. deep brain stimulation)
* With medication-resistant freezing of gait
* Significant cognitive impairment (Montreal Cognitive Assessment score <18)
* Unstable medical conditions
* Other neurological conditions
* Unable to follow instructions or safely complete the training tasks

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
General task performance (response time of the random sequence) at initial retention, adjusted for baseline | Day 8 (i.e. 48 hours after the last block of training)
  Response time of the random sequence within initial retention trial, adjusted for baseline (i.e. the first trial of acquisition on Day 3)
Implicit sequence learning (difference in response time between the random and repeated sequences) at initial retention, adjusted for baseline | Day 8 (i.e. 48 hours after the last block of training)
  The difference in response time between the random and repeated sequences of the initial retention trial, adjusted for baseline (i.e. the first trial of acquisition on Day 3)

SECONDARY OUTCOMES:
Immediate decrement (difference in response time between initial retention and the last trial of acquisition) in general task performance, adjusted for baseline | Day 5, Day 8 (i.e. 48 hours after the last block of training)
  The difference in response time of the random sequence within the initial retention trial and the last trial of acquisition, adjusted for baseline (i.e. first trial of acquisition)
Delayed decrement (difference in response time between delayed retention and the last trial of acquisition) in general task performance, adjusted for baseline | Day 5, Day 13-15 (i.e. at least 7 days after the last block of training)
  The difference in response time of the random sequence within the delayed retention trial and the last trial of acquisition, adjusted for baseline (i.e. first trial of acquisition)
Immediate decrement (difference in response time between initial retention and the last trial of acquisition) in implicit sequence learning (difference in response time between the random and repeated sequences), adjusted for baseline | Day 5, Day 8 (i.e. 48 hours after the last block of training)
  The difference in response time between the random and repeated sequences of the last trial of acquisition subtracted from the difference in response time between the random and repeated sequences of the initial retention trial, adjusted for baseline (i.e. first trial of acquisition)
Delayed decrement (difference in response time between delayed retention and the last trial of acquisition) in implicit sequence learning (difference in response time between the random and repeated sequences), adjusted for baseline | Day 5, Day 13-15 (i.e. at least 7 days after the last block of training)
  The difference in response time between the random and repeated sequences of the last trial of acquisition subtracted from the difference in response time between the random and repeated sequences of the delayed retention trial, adjusted for baseline (i.e. first trial of acquisition)
Four Square Step test score, adjusted for baseline | Day 13-15 (i.e. at least 7 days after the last block of training)
  Time taken to complete the Four Square Step test at delayed retention, adjusted for baseline (Four Square Step test score at baseline, i.e. 3 days prior to the first block of training)
MiniBEST score, adjusted for baseline | Day 13-15 (i.e. at least 7 days after the last block of training)
  MiniBEST score at delayed retention, adjusted for baseline (MiniBEST score at baseline, i.e. 3 days prior to the first block of training)

CONTACTS AND LOCATIONS:
Overall Officials: Serene S Paul, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States